CLINICAL TRIAL: NCT02115958
Title: Study of Cancer Stem Cell Vaccine That as a Specific Antigen in Metastatic of the Nasopharynx
Brief Title: The Immunotherapy of Nasopharyngeal Cancer Using Cancer Stem Cells Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLN-001; 201401 (Other Grant/Funding Number: The research fund of Fuda cancer hospital in Guangzhou)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2014-04

CONDITIONS: Neoplasms, Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- non-cancer stem cell vaccine (Placebo Comparator): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving low dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving middle dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving high dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine

INTERVENTIONS:
Biological: cancer stem cell vaccine

SUMMARY:
Most studies of cancer stem cells (CSC) involve the inoculation of cells from human tumors into immunosuppressed mice, preventing an assessment on the immunologic interactions and effects of CSCs. In this study, the investigators examined the vaccination effects produced by CSC-enriched populations from histologically distinct murine tumors after their inoculation into different syngeneic immunocompetent hosts. Enriched CSCs were immunogenic and more effective as an antigen source than unselected tumor cells in inducing protective antitumor immunity.Immune sera from CSC-vaccinated hosts contained high levels of IgG which bound to CSCs, resulting in CSC lysis in the presence of complement.CTLs generated from peripheral blood mononuclear cells or splenocytes harvested from CSC-vaccinated hosts were capable of killing CSCs in vitro. Mechanistic investigations established that CSC-primed antibodies and T cells were capable of selective targeting CSCs and conferring antitumor immunity.

DETAILED DESCRIPTION:
To assess the feasibility of generating CSC-loaded DC vaccines for clinical use, the investigators will harvest peripheral blood and tumor specimen from patients with Nasopharyngeal Cancer. The investigators will purify T, B cells and generate DCs from the PBMCs of the nasopharyngeal cancer patient.On the other hand, investigators will isolate ALDHhigh and ALDHlow tumor cells from the tumor specimen of the nasopharyngeal cancer patient using a similar protocol as investigators reported .

Aim 1: To demonstrate, in vitro, the relative cellular anti-nasopharyngeal cancer CSC immunity induced by nasopharyngeal cancer CSC-DC primed cytotoxic T cells.

Aim 2: To determine, in vitro, specific binding and lysis of nasopharyngeal cancer CSCs by antibodies produced by purified B cells from PBMCs stimulated with nasopharyngeal cancer CSC-DC.

ELIGIBILITY:
Inclusion Criteria:

* 1.patients are greater than 18 years of age, with advanced local disease (T3-T4N0-1M0), nodal disease (T1-T2N2-3M0) and loco-regional disease (T3-T4N2-3M0) at onset but presently controlled by standard therapy (combination of chemotherapy and radiotherapy) or with completely resected metastatic disease.

  2.Pathologic confirmation of nasopharyngeal carcinoma by the NCI Laboratory of Pathology (NPC).

  3.serum creatinine of 2.0 mg/dl or less. 4.Total bilirubin 1.6 mg/dl or less, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

  5.WBC 3000/mm(3) or greater. 6.platelet count 90,000 mm(3) or greater. 7.serum AST/ALT less than three times normal. 8.ECOG performance status of 0 or 1. 9.Patients of both genders must be willing to practice effective birth control during this trial because the potential for teratogenic effects are unknown.

  10.Patients may have had prior adjuvant treatment or may have had treatment for metastatic disease and are now with no evidence of disease, including chemotherapy or biotherapy, as long as 1 month has elapsed since prior systemic therapy.

Exclusion Criteria:

1. Patients who test positive for Hepatitis B virus, Hepatitis C virus or HIV. 2. level 3 hypertension; 3. severe coronary disease; 4. myelosuppression; 5. respiratory disease; 6. brain metastasis; 7. chronic infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The primary study purpose to determine the safety of immunization with cancer stem cells vaccine by the number of participants with adverse events | up to 3 months

SECONDARY OUTCOMES:
The secondary objectives are to evaluate vaccine immune responses to the immunizations by the data of body measurements | 1 month

OTHER OUTCOMES:
The dose of CSC vaccine | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Ning N, Pan Q, Zheng F, Teitz-Tennenbaum S, Egenti M, Yet J, Li M, Ginestier C, Wicha MS, Moyer JS, Prince ME, Xu Y, Zhang XL, Huang S, Chang AE, Li Q. Cancer stem cell vaccination confers significant antitumor immunity. Cancer Res. 2012 Apr 1;72(7):1853-64. doi: 10.1158/0008-5472.CAN-11-1400. PMID 22473314
- See also: Related Info — http://www.fudahospital.com/